CLINICAL TRIAL: NCT02644486
Title: A Prospective, Single-center, Randomized, Controlled Study of Sevelamer Carbonate in the Lipid Metabolism and Uric Acid Treatment of Obesity-Related Glomerulopathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty in enrollment
Sponsor: Zhi-Hong Liu, M.D. (Other)
Responsible Party: Sponsor-Investigator, Zhi-Hong Liu, M.D., professor, Nanjing University School of Medicine
Organization: Nanjing University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-1406
Record Dates: First submitted 2015-12-30; First posted 2015-12-31 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Obesity and Glomerulopathy
MeSH Terms: conditions — Obesity | interventions — Irbesartan

ARMS (3):
- A Group (Experimental)
  Interventions: Drug: High dosage Sevelamer Carbonate + Irbesartan
- B Group (Experimental)
  Interventions: Drug: Low dosage Sevelamer Carbonate + Irbesartan
- C Group (Active Comparator)
  Interventions: Drug: Irbesartan

INTERVENTIONS:
Drug: High dosage Sevelamer Carbonate + Irbesartan — Sevelamer Carbonate 4.8g/d+Irbesartan 300mg/d
  Arms: A Group
Drug: Low dosage Sevelamer Carbonate + Irbesartan — Sevelamer Carbonate 2.4g/d+Irbesartan 300mg/d
  Arms: B Group
Drug: Irbesartan — Irbesartan 300mg/d
  Arms: C Group

SUMMARY:
To observe the decreased levels of low-density lipoprotein from baseline in patients with obesity-related glomerulopathy (ORG) after 12 weeks of Sevelamer Carbonate treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of obesity
* diagnosed ORG by renal biopsy
* LDL>3.37mmol/L
* Proteinuria 0.5-3.5g/d
* eGFR (CKD-EPI formula) > 30ml/min

Exclusion Criteria:

* Other concomitant renal diseases
* Endocrine or drug-induced obesity;
* Type 2 diabetes
* eyes or obvious microscopic hematuria;
* Swallowing difficulty / severe gastrointestinal dysfunction
* intestinal obstruction;
* severe arrhythmia;
* Hypophosphatemia (<0.7mmol/L);
* allergic to Sevelamer Carbonate
* unable to well cooperate
* Females who are in the period of gestation or lactation, or refuse to use contraception;
* participated in other clinical trial of drug within three months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
low-density lipoprotein | 12 weeks
  decreased levels of low-density lipoprotein from baseline

SECONDARY OUTCOMES:
uric acid | 12 weeks
  Changes of uric acid from baseline after 12 weeks of treatment
blood lipids parameters (CHO, TG, HDL) | 12 weeks
  Changes of blood lipids parameters from baseline after 12 weeks of treatment
proteinuria | 12 weeks
  Changes of proteinuria from baseline after 12 weeks of treatment
blood glucose | 12 weeks
  Changes of blood glucose from baseline after 12 weeks of treatment
glycated hemoglobin | 12 weeks
  Changes of glycated hemoglobin from baseline after 12 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing, Jiangsu, China